CLINICAL TRIAL: NCT00082654
Title: Emotional Needs of Caregivers and Patient/Spouse Couples During Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Study of the Emotional Needs of Caregivers of Stem Cell Transplantation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 1639.00; CDR0000355106
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Neuroblastoma; Ovarian Cancer; Psychosocial Effects of Cancer and Its Treatment; Testicular Germ Cell Tumor
Keywords: psychosocial effects of cancer and its treatment; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative disease, unclassifiable; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III multiple myeloma; stage III ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV ovarian epithelial cancer; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Understanding the emotional needs of spouses or others who are living with and caring for patients who have undergone stem cell transplantation may help improve the quality of life of both the caregivers and the patients.

PURPOSE: This clinical trial is studying the emotional needs of caregivers of patients who have undergone stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess expression of emotion, as a function of patient presence, among spousal or other cohabiting caregivers (CG) of post-hematopoietic stem cell transplantation patients.
* Assess desynchrony among subjective (self-report) and expressive indicators of emotion, as a function of patient presence, in these participants.
* Correlate CG dispositional inhibition and desynchrony with physical and marital satisfaction in these participants.

OUTLINE: Caregivers (CG) complete written questionnaires assessing demographics, positive and negative affect, dispositional inhibition, marital satisfaction, and physical health over 45 minutes to 1 hour on day 1. CG then engage in two oral emotional expression exercises (on the topic of caregiving and the transplant) over 2 hours on day 2. Patients are present for one oral emotional expression exercise.

Participants are followed at 2 weeks and 6 months.

PROJECTED ACCRUAL: A total of 60 patient/spouse couples will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* In a marriage OR long-term, committed, heterosexual or homosexual, cohabiting relationship in which one member is post-hematopoietic stem cell transplantation

  * Patients must meet the following criteria:

    * At least 1 year since prior first bone marrow, stem cell, or umbilical cord blood transplantation

      * Allogeneic or autologous
    * Diagnosis of malignancy, myelodysplasia, or non-malignancy
    * No indication of possible or confirmed relapse
  * Spouse/caregiver (CG) must meet the following criteria:

    * Serve as the primary CG to the patient
    * No prior or concurrent neurologic disorder

PATIENT CHARACTERISTICS:

Age

* 21 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No concurrent major psychiatric disorder
* English-speaking

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Langer, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States